CLINICAL TRIAL: NCT07121686
Title: Effect of Red and Blue Light Irradiation on Wound Healing After Hemorrhoid Surgery: A Single - Center Prospective Open - Label Randomized Clinical Trial
Brief Title: Effect of Red and Blue Light Irradiation on Wound Healing After Hemorrhoid Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHPutianU 2024212-1
Record Dates: First submitted 2025-08-04; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: Control group:After internal haemorrhoid ligation + external haemorrhoidectomy, patients were given routine potassium permanganate sitz baths and routine nursing care to encourage patients to carry out functional exercises in moderation, mainly anal lifting, buttock lifting and abdominal massage.
  Red light group:Based on the control group, red light irradiation wound treatment was used; Red and blue light group: based on the control group, red and blue light irradiation trauma treatment was used;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Care Group (No Intervention): Standard postoperative care for hemorrhoidectomy patients.
- Red Light Therapy Group (Experimental): Conventional care plus red light phototherapy.
  Interventions: Device: Red light exposure
- Red-Blue Light Therapy Group (Experimental): Conventional care plus combined red-blue light phototherapy.
  Interventions: Device: Red-blue light exposure

INTERVENTIONS:
Device: Red light exposure — Patients in the red light group received red light therapy concurrently with standard care.
  Arms: Red Light Therapy Group
Device: Red-blue light exposure — Patients in the red and blue light group received combined red and blue light therapy concurrently with standard care.
  Arms: Red-Blue Light Therapy Group

SUMMARY:
The subjects of this study were patients who took mixed haemorrhoidectomy during the period of December 2024 - December 2025 . The haemorrhoidectomy patients were randomly divided into routine group, red light group and red and blue light group, and were given different ways of trauma care, and the number of cases in each group was 105 , with a total of 305 cases. Observe the difference between red and blue light irradiation and routine care on the healing time of postoperative trauma and postoperative complications after haemorrhoidectomy, and evaluate the patients' quality of life and satisfaction with treatment under both red light irradiation and routine care.

DETAILED DESCRIPTION:
The subjects of this study were patients who took mixed haemorrhoidectomy during the period of December 2024 - December 2025 . The diagnostic criteria were haemorrhoidal disease diagnosed as degree III-IV according to Goligher's classification. Inclusion criteria were 18 years < age < 75 years; diagnosis of haemorrhoids; internal haemorrhoid ligation + external haemorrhoidectomy. Exclusion criteria were patients with psychiatric disorders; patients with chronic diseases such as diabetes mellitus, hypertension and coronary artery disease; patients who underwent other treatments in addition to haemorrhoidectomy such as haemorrhoidal radiofrequency ablation/ sclerotherapy; patients who were unable to cooperate with the follow-up; and patients with perianal abscess, anal fissure, anal fistulae, and anorectal papillae hypertrophy. The haemorrhoidectomy patients were randomly divided into the conventional group, the red light group and the red and blue light group, and were given different ways of trauma care, and the number of cases in each group was 105 , with a total of 305 cases. The control group was given routine potassium permanganate sitz bath and routine care after internal haemorrhoid ligation + external haemorrhoidectomy to encourage patients to carry out functional exercise in moderation, mainly for anal lifting, buttock lifting and abdominal massage, etc.; the red light group was based on the control group, using red light irradiation for traumatic treatment; the red and blue light group was based on the control group, using red and blue light irradiation for traumatic treatment. Observe the difference between red and blue light irradiation and routine care on the healing time of postoperative trauma and postoperative complications after haemorrhoid surgery, and evaluate the patients' quality of life and satisfaction with treatment under both red light irradiation and routine care. Specific research content is to collect the postoperative data of the three groups of patients, including the recording of surgery-related pain scores, respectively, before the red light intervention and after the intervention of 1 d, 2 d, 3 d, 5 d, 7 d using visual analogue scoring (VAS) to assess the intensity of the patient's pain; the recording of the length of hospital stay; the recording of the degree of oedema of the anal verge were assessed before the red light intervention and after the intervention of 1 d, 2 d, 3 d, 5 d, 7 d, respectively, 0 Score 0: no oedema or slight oedema on the wound, but no impact on life. Score 2: oedema is present in only one area of the wound and is less than 1 cm in diameter, affecting daily activities. 4 points: multiple oedemas with a diameter of 1-2 cm, affecting daily activities. 6 points: multiple oedemas with a diameter of more than 2 cm, seriously affecting daily activities; follow up on the time to complete healing of the wound, quality of life scores, and the patient's satisfaction with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Diagnosed with Grade III-IV hemorrhoids according to Goligher classification
* Scheduled to undergo rubber band ligation of internal hemorrhoids + external hemorrhoidectomy
* Willing and able to provide written informed consent
* Able to comply with postoperative follow-up and treatment protocol

Exclusion Criteria:

* Psychiatric disorders or cognitive impairment
* Uncontrolled chronic diseases:
* Diabetes (HbA1c >7.5%)
* Hypertension (BP >160/100 mmHg)
* Coronary artery disease (NYHA Class III-IV heart failure)
* Concurrent other hemorrhoid treatments (e.g., radiofrequency ablation/sclerotherapy)
* Inability to complete follow-up (e.g., living too far away, no stable contact)
* Concurrent anal disorders:
* Perianal abscess
* Anal fissure
* Anal fistula
* Hypertrophied anal papilla
* Pregnancy or lactation (for female patients)
* History of phototherapy allergy
* Participation in other clinical trials within 3 months

For registration, simply copy this structured list directly into the PRS system's eligibility section. The clear formatting will facilitate efficient review.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | Daily from Day 1 until complete epithelialization (max 28 days post-op)
  Defined as 100% re-epithelialization assessed by blinded evaluator

SECONDARY OUTCOMES:
Postoperative pain intensity (VAS score) | Baseline, Day 1, 2, 3, 5, 7, and Day 14±2
  Assessed at rest and during defecation
Perianal edema severity (0-6 scale) | Day 1, 2, 3, 5, 7, and Day 14±2
  Evaluated by trained research nurses
Length of hospital stay | From surgery end to discharge (up to 7 days)
  Measured in hours with standardized discharge criteria
Complication incidence | Within 30 days postoperatively
  Classified by Clavien-Dindo grading system

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Putian University, Putian, China